CLINICAL TRIAL: NCT03394157
Title: Efficacy of Sleeve Gastrectomy, MGB, SASI Bypass in Type 2 Diabetes Obese Patients, Comparative Randomized Study
Brief Title: Randomized Comparative Study of Sleeve Gastrectomy Versus MGB and SASI Bypass , Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: tarek mahdy (Other)
Responsible Party: Sponsor-Investigator, tarek mahdy, professor of Bariatric and Metabolic surgery, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QGS1101
Record Dates: First submitted 2017-12-29; First posted 2018-01-09 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: sleeve gastrectomy , MGB , type 2 diabetes , obesity , SASI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes Mellitus Type 2 in Obese patients (Other): obese patients had metabolic surgery for the treatment for DMT2 .Preoperative data , which including SASI bypass , MGB and Sleeve gastrectomy
  Interventions: Other: metabolic surgery

INTERVENTIONS:
Other: metabolic surgery — operation to cure type2 diabetes
  Other Names: diabetic surgery

SUMMARY:
the investigator Randomized and compare the efficacy of 3 types of metabolic surgery in the treatment of type 2 diabetes in obese patients, one of them is SASI bypass which is a modification of Santoro's operation by performing a loop rather than Roux-en-Y bipartition reconstruction and the investigator are reporting the first comparative clinical trial as regards the clinical results of the outcomes of SASI bypass as a mode of functional restrictive and neuroendocrine modulation therapeutic option for obese type 2 diabetes.

DETAILED DESCRIPTION:
from 2011 to 2017, investigators Randomized and collect data for the 3 operations SASI bypass , Mini gastric bypass and Sleeve gastrectomy ) about thorough history, clinical examination and laboratory investigations including basic preoperative investigations, lipid profile, thyroid and suprarenal hormonal evaluation. In addition, patients may undergo further assessment for pulmonary functions or gastroesophageal disease including endoscope. . Abdominal ultrasound was done to exclude gall stones and to evaluate the degree of fatty liver. Reduction the size of fatty liver was done by putting all patients on low-calorie protein diet for 6 weeks. Deep vein thrombosis prophylaxis started 12 h before surgery with low molecular weight heparin subcutaneous injections . Preoperative data included age, gender, initial weight, initial body mass index (BMI), obesity complications and treatment medications used (chest problems, diabetes, arterial hypertension and cardiac ischaemia, hyperlipidemia, obstructive sleep apnea syndrome, gall stones, urinary stress incontinence, joint pain, depression, infertility and heart burn). Postoperative data included hospital stay, early postoperative complications during the first month (e.g. fever, collection, bleeding, vomiting, leak and port site problems .Long-term complications more than 1 month after surgery (e.g. nausea, vomiting, reflux, stricture, intestinal obstruction , hypoalbuminemia , anemia and calcium or iron or vitamin D , vitamin B12 deficiency and), excess weight loss and BMI were collected.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetic obese patients

Exclusion Criteria:

* patients age above 65 or below 18 years old
* history of upper laparotomy
* unfit for anesthesia or laparoscopy
* major psychological instability
* drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
excess weight loss | one year
  The percent of excess weight loss was calculated as follows: [(preoperative weight-follow up weight)/preoperative excess weight] ×100.

SECONDARY OUTCOMES:
Resolution of diabetes | one year
  defined in this study as a fasting plasma glucose level < 110 mg/dL or HbA1C level < 6 % without hypoglycemic medication at 1 year after surgery. whereas improvement was defined as a reduction of at least 25% in the fasting plasma glucose level and of at least 1% in the hemoglobin A1c level with hypoglycemic drug treatment

IPD SHARING:
Plan to Share IPD: Undecided